CLINICAL TRIAL: NCT03826888
Title: Measurement of Different Anti-Müllerian Hormone Isoforms in Expected Poor Responders: Does it Matter?
Brief Title: Measurement of Different Anti-Müllerian Hormone Isoforms in Expected Poor Responders
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Melado, IVF Specialist, ART Fertility Clinics LLC
Other Study IDs: 1807-ABU-055-LM
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Anti-Mullerian Hormone Isoforms
Keywords: IVF; AMH isoforms; ovarian reserve test; poor response

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study wants to evaluate significant clinical impact of different AMH isoforms in serum can be present or absent in expected poor responder participants. The specific AMH isoforms could therefore be measured in expected poor responder participants in order to obtain a more realistic clinical picture and therefore be able to give proper information to the participants and selection of medication dose for ovarian stimulation.

DETAILED DESCRIPTION:
The study has a prospective observational multicentric design and the investigators aim to investigate the presence of AMH isoforms and the levels of Inhibin B in serum among a population of participants with low ovarian reserve (AMH blood test below 1.1 ng/ml). Transvaginal scan for AFC and blood drawn from participants will be obtained on day 2-3 of menstrual period. The serum will be divided for AMH analysis using different assays: Elecsys Cobas assay for AMH and AnshLabs AMH isoforms specific assays (picoAMH 24/32 Pro-Mature, 24/37 Midpro-Midpro, 17/15 Mature-Mature and 10/24 Pro-Midpro) and AnshLabs Inhibin B ELISA.

Clinically it is not uncommon to see a discrepancy between the AFC count and the levels of AMH; this could be potentially explained by the presence of different AMH isoforms not measured with conventional commercial assays. Also, the evaluation of Inhibin B may be helpful for ovarian reserve assessment. Quantitation of specific Isoforms of AMH by different ELISA methods will investigate a possible relationship(s) between specific isoforms of AMH and poor responders.

ELIGIBILITY:
Inclusion Criteria:

* pre-treatment AMH recording below 1.1 ng/ml on day 2 or 3 of the menstrual cycle.
* BMI between 18 and 30 kg/m2.

Exclusion Criteria:

* Pregnancy.
* Breastfeeding.
* Intake of oral contraceptive pills or steroids for the last two menstrual cycles.
* Endometriosis.
* Previous surgical intervention, which could have an impact on the ovarian reserve, e.g. ovarian cyst removal, removal of one or both tubes, tubal ligation for sterilisation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Infertile female undergoing ovarian stimulation
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
AMH serum levels | 1 day
  Differences in AMH serum levels due to the presence of different AMH isoforms when results are compared with AMH measurement in blood performed with Elecsys Cobas AMH assay.

SECONDARY OUTCOMES:
Inhibin B and ovarian reserve markers | 1 day
  Correlation between Inhibin B and ovarian reserve markers (AMH serum levels and AFC)
AMH serum and AFC | 1 day
  Correlation between AMH serum levels (measured with different ELISA tests) and AFC.

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Middle East Fertility Clinic, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] McLennan IS, Pankhurst MW. Anti-Mullerian hormone is a gonadal cytokine with two circulating forms and cryptic actions. J Endocrinol. 2015 Sep;226(3):R45-57. doi: 10.1530/JOE-15-0206. Epub 2015 Jul 10. PMID 26163524
- [Background] Cate RL, Mattaliano RJ, Hession C, Tizard R, Farber NM, Cheung A, Ninfa EG, Frey AZ, Gash DJ, Chow EP, et al. Isolation of the bovine and human genes for Mullerian inhibiting substance and expression of the human gene in animal cells. Cell. 1986 Jun 6;45(5):685-98. doi: 10.1016/0092-8674(86)90783-x. PMID 3754790
- [Background] Josso N, Belville C, di Clemente N, Picard JY. AMH and AMH receptor defects in persistent Mullerian duct syndrome. Hum Reprod Update. 2005 Jul-Aug;11(4):351-6. doi: 10.1093/humupd/dmi014. Epub 2005 May 5. PMID 15878900
- [Background] Pankhurst MW, McLennan IS. Human blood contains both the uncleaved precursor of anti-Mullerian hormone and a complex of the NH2- and COOH-terminal peptides. Am J Physiol Endocrinol Metab. 2013 Nov 15;305(10):E1241-7. doi: 10.1152/ajpendo.00395.2013. Epub 2013 Sep 17. PMID 24045871
- [Background] Pankhurst MW, Chong YH, McLennan IS. Enzyme-linked immunosorbent assay measurements of antimullerian hormone (AMH) in human blood are a composite of the uncleaved and bioactive cleaved forms of AMH. Fertil Steril. 2014 Mar;101(3):846-50. doi: 10.1016/j.fertnstert.2013.12.009. Epub 2014 Jan 11. PMID 24424371
- [Background] Pankhurst MW, Clark CA, Zarek J, Laskin CA, McLennan IS. Changes in Circulating ProAMH and Total AMH during Healthy Pregnancy and Post-Partum: A Longitudinal Study. PLoS One. 2016 Sep 9;11(9):e0162509. doi: 10.1371/journal.pone.0162509. eCollection 2016. PMID 27612037
- [Background] Robertson DM, Kumar A, Kalra B, Shah S, Pruysers E, Vanden Brink H, Chizen D, Visser JA, Themmen AP, Baerwald A. Detection of serum antimullerian hormone in women approaching menopause using sensitive antimullerian hormone enzyme-linked immunosorbent assays. Menopause. 2014 Dec;21(12):1277-86. doi: 10.1097/GME.0000000000000244. PMID 24781853
- [Background] Robertson DM, Hale GE, Fraser IS, Hughes CL, Burger HG. Changes in serum antimullerian hormone levels across the ovulatory menstrual cycle in late reproductive age. Menopause. 2011 May;18(5):521-4. doi: 10.1097/gme.0b013e3181f8d9e0. PMID 21178792
- [Background] Gnoth C, Schuring AN, Friol K, Tigges J, Mallmann P, Godehardt E. Relevance of anti-Mullerian hormone measurement in a routine IVF program. Hum Reprod. 2008 Jun;23(6):1359-65. doi: 10.1093/humrep/den108. Epub 2008 Apr 2. PMID 18387961
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Kedem A, Haas J, Geva LL, Yerushalmi G, Gilboa Y, Kanety H, Hanochi M, Maman E, Hourvitz A. Ongoing pregnancy rates in women with low and extremely low AMH levels. A multivariate analysis of 769 cycles. PLoS One. 2013 Dec 16;8(12):e81629. doi: 10.1371/journal.pone.0081629. eCollection 2013. PMID 24363812
- [Background] Koshy AK, Gudi A, Shah A, Bhide P, Timms P, Homburg R. Pregnancy prognosis in women with anti-Mullerian hormone below the tenth percentile. Gynecol Endocrinol. 2013 Jul;29(7):662-5. doi: 10.3109/09513590.2013.797395. PMID 23772777
- [Background] Seifer DB, Tal O, Wantman E, Edul P, Baker VL. Prognostic indicators of assisted reproduction technology outcomes of cycles with ultralow serum antimullerian hormone: a multivariate analysis of over 5,000 autologous cycles from the Society for Assisted Reproductive Technology Clinic Outcome Reporting System database for 2012-2013. Fertil Steril. 2016 Feb;105(2):385-93.e3. doi: 10.1016/j.fertnstert.2015.10.004. Epub 2015 Oct 26. PMID 26515380
- [Background] Broekmans FJ, de Ziegler D, Howles CM, Gougeon A, Trew G, Olivennes F. The antral follicle count: practical recommendations for better standardization. Fertil Steril. 2010 Aug;94(3):1044-51. doi: 10.1016/j.fertnstert.2009.04.040. Epub 2009 Jul 8. PMID 19589513
- [Derived] Melado L, Kumar A, Kalra B, Kalafat E, Lawrenz B, Fatemi H. How to enhance prediction of clinical outcomes in poor responders: integrating high-specific assays for anti-mullerian hormone with antral follicle count. Front Endocrinol (Lausanne). 2025 Sep 29;16:1654365. doi: 10.3389/fendo.2025.1654365. eCollection 2025. PMID 41089290
- [Derived] Melado L, Kumar A, Kalra B, Kalafat E, Lawrenz B, Fatemi H. The role of bioavailable inhibin B in predicting oocyte yield in expected poor responders: the forgotten marker? J Assist Reprod Genet. 2025 Nov;42(11):3913-3920. doi: 10.1007/s10815-025-03637-9. Epub 2025 Aug 27. PMID 40866738